CLINICAL TRIAL: NCT03144050
Title: Optical Imaging For Assessment of Foot Perfusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Modulated Imaging Inc. (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 11150
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Ulcer Foot; Diabetes
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 0: Control - no diabetes
  Interventions: Device: SFDI Imaging
- 1: Diabetes
  Interventions: Device: SFDI Imaging
- 2: Diabetes w/neuropathy
  Interventions: Device: SFDI Imaging
- 3: Diabetes with vascular disease
  Interventions: Device: SFDI Imaging
- 4: Diabetes w/healed ulcer
  Interventions: Device: SFDI Imaging
- 5: Diabetes with current ulcer
  Interventions: Device: SFDI Imaging

INTERVENTIONS:
Device: SFDI Imaging — Imaging with SFDI device
  Other Names: OxImager

SUMMARY:
This study is designed to evaluate the ability of Spatial Frequency Domain Imaging (SFDI) to measure perfusion in lower extremities and to understand how it might be used in a podiatry clinic.

DETAILED DESCRIPTION:
This study is designed to evaluate the ability of Spatial Frequency Domain Imaging (SFDI) to measure perfusion in lower extremities and to understand how it might be used in a podiatry clinic. SFDI is a non-contact optical imaging technology that measures tissue functional (blood volume, tissue oxygen saturation) and structural information (scattering index) across a large field of view. Our hypothesis is that SFDI parameters can eventually become a quantitative tool to assess foot health and identify patients at risk for ulcer formation. This phase of the study is designed to correlate SFDI outputs to current clinical risk categories

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Pregnant/lactating women
* Rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any person at risk for foot ulcer formation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-07-31 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical risk category | immediate
  risk assessment based on clinical signs

SECONDARY OUTCOMES:
Ulcer incidence | 1 year
  Ulcer formation

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided